CLINICAL TRIAL: NCT02516033
Title: Identification of a Risk Profile Associated With Failure of the Hybrid Ablation of Atrial Fibrillation.
Brief Title: Hybrid Atrial Fibrillation Ablation Registry
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, I.C. Van Gelder, prof., University Medical Center Groningen
Other Study IDs: METc2014/239
Record Dates: First submitted 2015-08-03; First posted 2015-08-05 (Estimated); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Hybrid Ablation; Efficacy; Risk Profile; Biomarkers
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Full blood sample
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Recently a combined approach of surgeon ablation in combination with endocardial ablation (hybrid ablation) has been introduced. This therapy has shown excellent results in patients with previous failed endocardial ablation for paroxysmal atrial fibrillation as well in patients with persistent atrial fibrillation. The investigators hypothesize that the severity of atrial remodeling in patients with atrial fibrillation can be measured by clinical factors, echocardiographic parameters, circulating biomarkers and genetic background, and that these factors can be used to identify a risk profile to predict failure of the hybrid ablation therapy in patients with atrial fibrillation. Aim of this study is to determine a risk profile based on clinical correlates, circulating biomarkers, and genetic background associated with failure of the hybrid ablation procedure, in a prospective single center registry setting. The investigators evaluate all consecutive patients who have agreed to undergo the hybrid ablation procedure because of atrial fibrillation. The investigators aim for a total of 250 participants. Extra study related procedures include blood sampling for biomarkers and genetic analysis, prolonged Holter monitoring for documentation of recurrences of atrial fibrillation/atrial flutter/atrial tachycardias, and a quality of life questionnaire. Total follow-up will be five years.

Main study endpoint is failure of the hybrid ablation procedure in patients with atrial fibrillation, i.e. any (a)symptomatic atrial fibrillation/atrial flutter/atrial tachycardia >30sec without anti-arrhythmic drugs at one year of follow-up by ECG recording and 3-day Holter monitoring.

DETAILED DESCRIPTION:
Rationale: The investigators hypothesize that the severity of atrial remodeling in patients with atrial fibrillation can be measured by clinical factors, echocardiographic parameters, circulating biomarkers and genetic background, and that these factors can be used to identify a risk profile to predict failure of the hybrid ablation therapy in patients with atrial fibrillation.

Objective: To determine a risk profile based on clinical correlates, circulating biomarkers, and genetic background associated with failure of the hybrid ablation procedure in patients with atrial fibrillation.

Study design: A prospective single center registry. Study population: Patients who have agreed to undergo the hybrid ablation procedure because of atrial fibrillation. The investigators aim for a total of 250 participants.

Intervention: Extra study related procedures include blood sampling for biomarkers and genetic analysis at baseline and 1 year follow-up; prolonged Holter monitoring for documentation of recurrences of atrial fibrillation/ atrial flutter/atrial tachycardias at 3 months, 6 months and 1 year follow-up; and a quality of life questionnaire at baseline, and at 1 year and 5 year follow-up.

Total follow-up duration: Five years. Main study endpoints: Failure of the hybrid ablation procedure in patients with atrial fibrillation, i.e. any (a)symptomatic atrial fibrillation/atrial flutter/atrial tachycardia >30sec without anti-arrhythmic drugs at one year of follow-up by ECG recording and 3-day Holter monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have agreed to undergo the hybrid ablation procedure because of atrial fibrillation.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have agreed to undergo the hybrid ablation procedure because of atrial fibrillation.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2015-01; Primary Completion 2024-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Failure of the hybrid ablation procedure in patients with atrial fibrillation | 1 year
  Any (a)symptomatic atrial fibrillation/atrial flutter/atrial tachycardia >30sec without anti-arrhythmic drugs at 1 year by ECG recording and 3-day Holter monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle C Van gelder, MD, PhD, Principal Investigator — University Medical Center Groningen

REFERENCES:
- [Derived] Velt MJH, Magni FT, Blaauw Y, Mariani MA, Klinkenberg TJ, Rienstra M, Mulder BA. Hybrid Atrial Fibrillation Ablation: Association of Clinical Characteristics, Biomarkers, and Blanking Period with Recurrence. Interdiscip Cardiovasc Thorac Surg. 2025 Sep 1;40(9):ivaf197. doi: 10.1093/icvts/ivaf197. PMID 40828897